CLINICAL TRIAL: NCT07236736
Title: Evaluation of SPM™ Topical Cosmetic Application on Skin Appearance, Hydration, and Barrier Support in Healthy Adults
Acronym: SPMT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biocoz Global Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1401971
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Healthy Skin; Skin Hydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPM™ Application Area (Experimental): Participants will apply the SPM™ topical cosmetic formulation twice daily for six (6) weeks to a designated skin area (e.g., right arm). SPM™ is a peptide-based cosmetic formulation containing amino acids, vitamins, and recombinant human serum albumin, designed to support healthy skin appearance, hydration, and barrier function.
  A matching contralateral site (e.g., left arm) will remain untreated and serve as the within-subject control for comparison. No product will be applied to this area.
  Skin biopsies (3-6 mm) will be obtained from both the treated and untreated sites at two timepoints:
  Baseline (before starting SPM™ application), and
  End of the 6-week product-use period.
  Biopsy samples from both sites will be analyzed in parallel to characterize cosmetic skin attributes (e.g., structure, hydration-related markers, and barrier-related characteristics) and to compare changes between the SPM™-treated and untreated control areas.
  Interventions: Procedure: Skin biopsy; Other: Corneometer® Measurement; Other: Tewameter® Measurement

INTERVENTIONS:
Procedure: Skin biopsy — Skin biopsies (3-6 mm) will be performed at two time points:
  Baseline (prior to initiation of SPM™ application)
  End of product-use period (after 6 weeks of twice-daily application)
  These samples will be analyzed for cosmetic-related skin structure and protein expression characteristics (e.g., filaggrin levels and barrier markers).
Other: Corneometer® Measurement — Noninvasive skin hydration assessment using the Corneometer® instrument at baseline and after 6 weeks. The device quantifies the moisture content of the stratum corneum through dielectric constant measurement.
Other: Tewameter® Measurement — Noninvasive transepidermal water loss (TEWL) measurement using the Tewameter® device to assess barrier function before and after the 6-week product-use period.

SUMMARY:
This is an exploratory, cosmetic-use study evaluating the effects of Super Protein Multifunction (SPM™), a topical peptide-based formulation, on skin appearance, hydration, and barrier-related characteristics in healthy adults. The study aims to collect preliminary biophysical and histologic data on cosmetic skin changes following six weeks of SPM™ use. Participants will apply the product to a designated skin area while a matched contralateral area serves as the untreated comparison site. Skin hydration, transepidermal water loss (TEWL), and tissue markers of skin structure and barrier integrity will be assessed before and after product use. The study includes noninvasive measurements and small punch biopsies at two timepoints.

DETAILED DESCRIPTION:
SPM™ is a multi-component peptide formulation designed to support skin health and barrier function. Preclinical data demonstrate reduced expression of inflammatory cytokines and potential improvements in epidermal physiology. Prior clinical data in eczematous skin suggest reductions in inflammation and improvements in clinician-assessed skin ratings. This pilot study extends investigation into healthy adults to characterize cosmetic and structural skin attributes associated with SPM™ use.

Participants aged 20-75 years will undergo screening, informed consent, and baseline assessments. Study procedures include Corneometer® hydration measurements, Tewameter® TEWL assessments, clinical photography, and 3-6 mm punch biopsies from both the application and comparison sites at baseline and end-of-treatment. Participants will apply SPM™ twice daily for 42 days. Follow-up phone calls occur after each biopsy to assess healing. A final safety follow-up visit occurs at Day 49 (±7 days) to evaluate recovery and participant-reported outcomes.

Biopsy samples will be analyzed at Mayo Clinic Pathology Core Laboratories to assess filaggrin expression and general histologic features. Additional exploratory biomarkers may be assessed in future IRB-approved studies using stored tissue.

Safety monitoring includes documentation of adverse events, with predefined stopping rules related to local tolerability, unexpected histologic findings, or systemic events. All study activities comply with ethical and regulatory standards, including 45 CFR 46, GCP, HIPAA, and WCG IRB oversight.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy with no systemic or active dermatologic diseases.
2. Willing and able to apply topical product daily for 6 weeks.
3. Able to provide written informed consent.
4. Willing to undergo skin biopsies and follow study procedures.

Exclusion Criteria:

1. History of skin cancer or other malignancy within the past 10 years.
2. Active or chronic dermatologic conditions (e.g., eczema, psoriasis, acne, rosacea).
3. Known allergy or sensitivity to components of the investigational product.
4. Current use of systemic corticosteroids or immunosuppressants.
5. Pregnancy or breastfeeding.
6. Any condition that, in the investigator's opinion, would interfere with study participation or pose additional risk.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-12-05 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in skin structure and protein expression (filaggrin levels) after 6 weeks of SPM™ topical application | Baseline (Day 0) and Week 6 - End of Product Use (Day 42 ± 7 days)
  To evaluate histologic and protein expression changes in skin tissue following six weeks of twice-daily SPM™ topical application, compared to baseline and to the untreated control area. Paired punch biopsies (3-6 mm) will be collected at baseline and after completion of product use. Filaggrin expression and general tissue features (e.g., epidermal thickness, keratinocyte morphology, and barrier integrity) will be assessed via immunohistochemistry and histologic analysis.

SECONDARY OUTCOMES:
Change in Skin Hydration | Baseline (Day 0) and Week 6 - End of Product Use (Day 42 ± 7 days)
  Skin hydration will be quantified using a Corneometer® device at baseline and after six weeks of product use. Measurements will be performed on both the SPM™-treated area and the contralateral untreated control area.
Change in Transepidermal Water Loss (TEWL) | Baseline (Day 0) and Week 6 - End of Product Use (Day 42 ± 7 days)
  Skin barrier function will be evaluated using a Tewameter® device to measure transepidermal water loss (TEWL) at baseline and after six weeks. Assessments will be performed at both treated and untreated areas to determine barrier-related effects of SPM™.
Change in Skin Appearance (Photographic Assessment) | Baseline (Day 0) and Week 6 - End of Product Use (Day 42 ± 7 days)
  Standardized clinical photographs will be captured under consistent lighting and positioning conditions at baseline and after six weeks to document visible changes in skin texture, tone, and smoothness. Images will be assessed for cosmetic improvements using qualitative scoring.
Safety and Tolerability (Adverse Events and Local Reactions) | Baseline (Day 0) and Week 6 - End of Product Use (Day 42 ± 7 days)
  Frequency and severity of product-related local skin reactions (e.g., erythema, irritation, dryness) and biopsy-related adverse events will be recorded and summarized.
Treatment Satisfaction Questionnaire for Medication 9 (TSQM-9). | End of study (Day 42-49)
  Participants will complete a self-reported questionnaire assessing perceived changes in skin comfort, hydration, smoothness, and overall cosmetic benefit after SPM™ use. Scores for each domain range from 0 to 100, with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Project Quality of Life, West Hollywood, California, United States